CLINICAL TRIAL: NCT01179841
Title: A Comprehensive Approach to Intervention for Toddlers at Risk for ASD
Brief Title: Intervention for Toddlers at Risk for Autism Spectrum Disorders (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Rebecca Landa, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00006553
Record Dates: First submitted 2010-07-21; First posted 2010-08-11 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; language; social; toddlers
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Playgroup and Parent Training (Experimental): 1. One to two-hour individual therapeutic sessions with parent training in the home or clinic, 1x every week over six months;
  2. parent training/enrichment once a week in our clinic for 20 sessions at 1-2 hours;
  3. a playgroup session for 1-2 hours 2x week for 6 months in our clinic and
  4. Community treatment as usual.
  Interventions: Behavioral: Playgroup; Behavioral: Parent Training
- Parent Training (Active Comparator): 1. Parent enrichment sessions once a week for 20 sessions (for 1-2 hours)
  2. Community treatment as usual.
  Interventions: Behavioral: Parent Training

INTERVENTIONS:
Behavioral: Playgroup — The playgroup will be conducted at our center and focuses on providing an invigorating learning environment in which emerging skills/knowledge are skillfully brought to a higher level of maturity, integrated with existing abilities, and used functionally. Learning with and through peers, provides the opportunity to address abnormal peer relationships for developmental level. Providing an enriched environment with toys, structured learning, and opportunities for ongoing engagement we offer the children experiences that they would not otherwise have. Parent training sessions will focus on strategies aimed at improving child social engagement and communication. Parent education sessions will focus on topics related to autism, learning styles, interventions, and resources.
  Arms: Playgroup and Parent Training
Behavioral: Parent Training — The 1-2 hour individual therapeutic sessions with parent training in the home or clinic (1x every week over six months) are based on our own program which is in development. This program focuses on teaching parents how to encourage social and communication skills in their toddlers and also provides comprehensive information about development. Sessions will focus on knowledge of autism, current access to services, general knowledge of strategies used to facilitate child development, advocacy, knowledge of how to access services, and coping strategies.
  Other Names: Enrichment Sessions
Behavioral: Parent Training — In the once-a-week 1 to 2 hour parent training/enrichment, we will ask parents to target specific play and care routines in which they may stimulate their child's development in the ways identified by the therapist. These stimulation times may be provided by the parents, other family members, friends, volunteers or hired assistants. Parents will be encouraged to have their child in direct skill-enhancing engagement for 1-2 hour per day. The therapist will work with the family to identify times during the day that best lend themselves to accomplishing this goal.
  Other Names: Individual Therapeutic Sessions
  Arms: Playgroup and Parent Training

SUMMARY:
This research is being done to test the effectiveness of an early intervention model for very young children at high risk for autism spectrum disorders (ASD) and their families. If children show improvement in this intervention, the investigators hope that the availability of public services of this type will be increased. Children between 11 months and 21 months old with Autism Spectrum Disorders, or with social and communication delays that indicate high risk for Autism Spectrum Disorders, and their parents may join the study. Treatment must start prior to the second birthday.

ELIGIBILITY:
Inclusion Criteria:

* Children will be ascertained between 11 months and 21 months of age
* Must be able to enter the study prior to their second birthday
* Must then pass an eligibility assessment to determine whether the child meets criteria for ASD and thus qualifies for the study. This assessment will consist of the Baby ADOS and the Mullen Scales of Early Learning. Children must meet criteria for ASD or autism on the ADOS, score more than one standard deviation below the mean on the Receptive or Expressive Language scale of the MSEL, and have a clinical judgment of ASD to be eligible for enrollment into treatment.
* Parents must agree to participate in the study and commit to having their child participate in the intervention to which they are randomized for 6 months
* The parent (or other primary caregiver, such as grandparent) in the Parent Enrichment/Training condition must agree to attend the training sessions

Exclusion Criteria:

* Fail hearing or vision screening (by pediatrician's office, audiologist, or ophthalmologist)
* Family's first language being other than English (language measures are normed on English speakers, putting non-English speakers at a disadvantage. In addition, the treatment is delivered in English. Children from non-English speaking homes may not make progress, but for reasons other than the efficacy of the intervention.)
* Head injury (because this may cause some of the symptoms, which may not be due to autism and therefore we would not be able to assess the effects of the intervention on autism)
* Identified reason for the autism (e.g., fragile X syndrome, Rett syndrome, Tuberous Sclerosis)
* Inability of the family to attend the playgroup sessions and parent trainings
* Parents whose hearing or vision is not within normal limits after correction (e.g., hearing aid, glasses)
* Parents with developmental delays, language or learning impairments, or a psychiatric diagnosis IF the impairment would interfere with parent training (PI will assess on a case by case basis by talking to the parent)
* Foster children
* Refusal to allow videotaping of the children's assessments or intervention or to allow videotaped footage to be used for teaching purposes.

Ages: 11 Months to 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Developmental Level | 3 months into treatment, 6 months into treatment, and 6 months after treatment ends
  Using the Mullen Scales of Early Learning to assess.

SECONDARY OUTCOMES:
Communication | 3 months after treatment starts
  Using Communication and Symbolic Behavior Scales to assess.
Communication | 6 months into treatment
  Using Communication and Symbolic Behavior Scales to assess.
Communication | 6 months after treatment ends
  Using Communication and Symbolic Behavior Scales to assess.
Presence and Severity of Autism | 3 months after treatment starts
  Using Autism Diagnostic Observation Schedule to assess.
Presence and Severity of Autism | 6 months into treatment
  Using Autism Diagnostic Observation Schedule to assess.
Presence and Severity of Autism | 6 months after treatment ends
  Using Autism Diagnostic Observation Schedule to assess.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Keen D, Rodger S, Doussin K, Braithwaite M. A pilot study of the effects of a social-pragmatic intervention on the communication and symbolic play of children with autism. Autism. 2007 Jan;11(1):63-71. doi: 10.1177/1362361307070901. PMID 17175574
- [Background] Solomon R, Necheles J, Ferch C, Bruckman D. Pilot study of a parent training program for young children with autism: the PLAY Project Home Consultation program. Autism. 2007 May;11(3):205-24. doi: 10.1177/1362361307076842. PMID 17478575
- [Background] Howlin P, Gordon RK, Pasco G, Wade A, Charman T. The effectiveness of Picture Exchange Communication System (PECS) training for teachers of children with autism: a pragmatic, group randomised controlled trial. J Child Psychol Psychiatry. 2007 May;48(5):473-81. doi: 10.1111/j.1469-7610.2006.01707.x. PMID 17501728